CLINICAL TRIAL: NCT03524534
Title: The Heart Failure Readmission Intervention by Variable Early Follow-up (THRIVE) Study
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: The Permanente Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CN-16-2667
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Follow-Up Intervention (Active Comparator)
  Interventions: Other: Telephone Call
- In-person follow-up intervention (Active Comparator)
  Interventions: Other: In-Person Primary Care Clinical Follow-Up Visit

INTERVENTIONS:
Other: Telephone Call — A phone call will take place within 7 days of discharge by a Kaiser Permanente Heart Failure Care Manager from the Kaiser Permanente Heart Failure Chronic Care Management Program.
  Arms: Telephone Follow-Up Intervention
Other: In-Person Primary Care Clinical Follow-Up Visit — This will be a standard in-person clinic visit with the subject's primary care physician within 7 days of discharge, with no structured heart failure protocol.
  Arms: In-person follow-up intervention

SUMMARY:
This study is a pragmatic randomized clinical trial to determine the effectiveness of two strategies of early follow-up in adults after hospitalization for heart failure: telephone follow-up with a heart failure care manager vs. in-person clinic visit with their primary care provider. The primary outcomes during 30-day follow-up will include readmission for heart failure, death and readmission for any cause. The study team aims to randomly assign 2400 patients during a 15-month period in a 1-to-1 ratio to either an initial structured telephone call with a heart failure care manager or an in-person primary care clinic visit within 7 days of discharge. A secondary goal is to increase the rate of any follow-up within 7 days of discharge to greater than 90 percent among all eligible patients.

DETAILED DESCRIPTION:
Heart failure (HF) affects >5 million adults nationally and is the leading cause of hospitalization among Medicare beneficiaries. Reducing hospitalization for heart failure (HF) and subsequent readmissions shortly after discharge is a nationally recognized health care delivery system priority. More than 20% of Medicare patients hospitalized for HF are readmitted within 30 days and this rate has not been declining over the past decade despite increasing attention to this problem. The data that will be collected could allow the study team to tailor the post-discharge follow-up program to patient characteristics to further improve the effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients hospitalized for confirmed acute heart failure at a Kaiser Permanente Northern California medical center

Exclusion Criteria:

* Planned discharge to a location other than their home. This includes a skilled nursing facility, nursing home or hospice facility.
* Planned discharge to home with hospice care.
* End-stage renal disease treated with chronic peritoneal dialysis or hemodialysis.
* Death during the index hospitalization.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2091 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Readmission for heart failure within 30-days | 30 days after discharge
  To compare 30-day rates of heart failure-related readmission for subjects randomly assigned to initial heart failure care manager telephone visit vs. in-person primary care clinic visit within 7 days after discharge from a heart failure hospitalization.

SECONDARY OUTCOMES:
Readmission for any cause within 30 days | 30 days after discharge
  To compare 30-day rates of readmission for any cause for subjects randomly assigned to initial heart failure care manager telephone visit vs. in-person primary care clinic visit within 7 days after discharge from a heart failure hospitalization.
Increase in 7-day follow-up rates | 7 days after discharge
  To increase follow-up rate within 7 days of discharge to > 90% in eligible patients
Death from any cause within 30 days | 30 days after discharge
  To compare 30-day rates of death from any cause for subjects randomly assigned to initial heart failure care manager telephone visit vs. in-person primary care clinic visit within 7 days after discharge from a heart failure hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Go, MD, Principal Investigator — Kaiser Permanente

REFERENCES:
- [Derived] Lee KK, Thomas RC, Tan TC, Leong TK, Steimle A, Go AS. The Heart Failure Readmission Intervention by Variable Early Follow-up (THRIVE) Study: A Pragmatic Randomized Trial. Circ Cardiovasc Qual Outcomes. 2020 Oct;13(10):e006553. doi: 10.1161/CIRCOUTCOMES.120.006553. Epub 2020 Sep 24. PMID 32967439